CLINICAL TRIAL: NCT02768376
Title: Spinal for Laparoscopic Cholecystectomy
Acronym: Sp-Lap
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, AlRefaey Kandeel, Dr, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Refa32016
Record Dates: First submitted 2016-05-03; First posted 2016-05-11 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Laparoscopic Cholecystectomy
MeSH Terms: interventions — Bupivacaine; Fentanyl; Anesthesia, Spinal; Injections, Spinal; Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- General anesthesia group (Active Comparator): General anesthesia group: Standard anesthetic technique will be applied.Anesthesia will be induced by propofol 1% (1-2 mg/kg), Fentanyl 1-2 mic/kg, and Atracurium 0.5 mg/kg then according to train of four response. Then maintained using Sevoflurane based anesthesia aiming to maintain Bispectral index 40-60..
  Interventions: Drug: General anesthesia
- Spinal anesthesia group (Experimental): While in sitting position; intrathecal injection using 25 G spinal needle using 3 mls of Bupivacaine 0.5% with 20 mic Fentanyl, at L 2-3 level the patient head will be lowered till sensory blockade of T6 obtained at least.
  Interventions: Drug: Bupivacaine with Fentanyl (Spinal Anesthesia)

INTERVENTIONS:
Drug: Bupivacaine with Fentanyl (Spinal Anesthesia) — Intrathecal injection of 15 mg Bupivacaine 0.5% at L 2-3 level mixed with 20 µ Fentanyl. Patients head will be lowered till sensory level of T 6 is abstained.
  Other Names: intrathecal
  Arms: Spinal anesthesia group
Drug: General anesthesia — Induction by propofl 1.5-2 mg/kg, Fentanyl 1-2 mic/kg and atracrium 0.5 mg/kg Then maintained using Sevoflurane based anesthesia aiming to maintain Bispectral index 40-60..
  Arms: General anesthesia group

SUMMARY:
In this study, the investigators will study spinal anesthesia for laparoscopic cholecystectomy in comparison to general anesthesia (GA) regarding patient satisfaction as a primary variable, intraoperative complications, postoperative analgesic requirements, postoperative nausea and vomiting, patient hospital stay (secondary variables).

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for laparoscopic cholecystectomy

Exclusion Criteria:

* coagulopathy
* Patient refusal
* previous spine surgery
* Obesity BMI more than 30

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-06 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction (over a scale from 1 to 4) | 24 hours
Postoperative analgesic consumption (mg morphine) | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university, Al Mansurah, Dkahleya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided